CLINICAL TRIAL: NCT04364334
Title: Collecting Diagnostic, Treatment and Follow-up Data on Knee Treatments.
Brief Title: Knee Registry (Knieregister)
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, R.J.H. Custers, Principal Investigator, UMC Utrecht
Other Study IDs: 17-005
Record Dates: First submitted 2020-04-15; First posted 2020-04-28 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Knee Pathology; Osteoarthritis, Knee; Osteochondritis Dissecans; Chondral Defect; Osteochondral Defect
Keywords: Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee registry patients

SUMMARY:
Rationale: In view of patient care, patient characteristics and treatment parameters are registered for all patients visiting the Mobility Clinic of the University Medical Center Utrecht for orthopaedic knee treatment. Patients also fill out questionnaires for function, pain and mobility of the knee, before and after treatment.

Objective: The main objective of this registry is to collect patient characteristics and treatment parameters together with data from the questionnaires in a database. This knee registry can be used for future research questions.

Study design: This is a longitudinal observational registry.

Study population: All patients that visit the Mobility Clinic will be asked to participate in the knee registry. Patients that meet one or more of the following criteria will be excluded: are below the age of 16, not able or willing to sign the broad consent form, not being able to read and understand Dutch language, or receiving medical treatment for their knee elsewhere.

Main study parameters/endpoints: Data will be collected for future research for which the purpose is not known at this time. When new research will be conducted, study parameters will be set. A study application has to be submitted to the institutional ethical review board of the University Medical Center Utrecht. Patients do not need to be asked permission for the use of their data for each study individually. Only when additional information is needed.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden for patients to participate in this registry is minimal and consists of time. Any future results may be beneficial for patients. Participation or refusal to participate in the registry has no consequences for their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Receives orthopaedic knee surgery or conservative knee treatment (advice, physiotherapy, injections etc) at the UMC Utrecht;
* Able to read and understand Dutch language;
* Is able and willing to signs the broad consent form.

Exclusion Criteria:

* Receives no treatment (refusal of surgery or treatment);
* Receives treatment elsewhere.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that visit the Mobility Clinic at the UMC Utrecht for their knee pathology.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2100-01 (Estimated); Study Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Patient characteristics and medical data | Status at baseline.
  General patient characteristics, medical data, and specific knee data.
Change in EQ5D (EuroQol 5 dimensions) | Before treatment, and after treatment at 3, 6, 9 (only for ACI patients) and 12 months. Then annually up to 20 years.
  The EQ-5D-5L is a questionnaire about the quality of life on a scale of 0-100 and has 5 dimensions, each dimension has 5 levels. A higher score indicates a higher health utility. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Change in KOOS (Knee Injury and Osteoarthritis Outcome Score) | Before treatment, and after treatment at 3, 6, 9 (only for ACI patients) and 12 months. Then annually up to 20 years.
  Questionnaire for evaluating limitations and symptoms for patients with knee complaints. Scale of 0-100, where 100 indicates no symptoms and limitations and 0 an extreme amount of symptoms and limitations.
Change in IKDC (International Knee Documentation Committee) | Before treatment, and after treatment at 3, 6 and 12 months. Then annually up to 20 years.
  Questionnaire about symptoms and function for patients with knee complaints. Scale of 0-100 where 100 indicates the highest level of function and lowest level of symptoms.
Change in SF-36 | Before treatment, and after treatment at 3, 6 and 12 months. Then annually up to 20 years.
  Questionnaire about the health related quality of life. There are several subcategories on a scale of 0-100, where a higher score indicates a better health related quality of life.
Change in VAS pain (Visual Analogue Scale) | Before treatment, and after treatment at 3, 6 and 12 months. Then annually up to 20 years.
  Question about pain on on a horizontal visual analogue scale, where the endpoints are labelled 'no pain' and 'unbearable pain'. This is converted into a scale of 0-100 where a higher score indicates a higher level of pain.
Change in NRS pain (Numeric Rating Scale) | Before treatment, and after treatment at 3, 6, 9 (only for ACI patients) and 12 months. Then annually up to 20 years.
  Question about the pain on a scale of 0 to 10 during rest and activity. 0 indicating no pain, 10 indicating extreme pain.
Change in Tegner | Before treatment, and after treatment at 3, 6 and 12 months. Then annually up to 20 years.
  Question about the level of work and sports activity on a scale from 0 to 10, where 10 indicates a high level of activity.
Anker questions | After treatment at 3, 6 and 12 months
  Questions about the results of surgery for functionality, pain and satifaction. Descriptive.
Change in OKS (Oxford knee score) | Before treatment, and after treatment at 3, 6 and 12 months. Then annually up to 20 years.
  Questionnaire about the pain and limitations of activities for patients with a knee prosthesis. Maximal total score is 60, indicating the maximum level of pain or functional limitations.
Change in healthcare use and costs | Before treatment, and after treatment at 6, 9 (only for ACI patients) and 12 months.
  iMTA-questionnaire descriptive (Medical Consumption and Productivity Cost Questionnaire)
Change in KOOS-PS (Knee Injury and Osteoarthritis Outcome Score-short form) | Before treatment, and after treatment at 3, 6 and 12 months. Then annually up to 20 years.
  Short form of the questionnaire for evaluating limitations and symptoms for patients with knee complaints. Scale of 0-100, where 100 indicates no symptoms and limitations and 0 an extreme amount of symptoms and limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Roel Custers, Dr, Principal Investigator — Orthopedic surgeon
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
New research questions that requires data from the registry need to be discussed and approved by the PI and data manager/coordinator of this registry. The proposal should also be in agreement with the research collaboration and data transfer guidelines and agreements of the UMC Utrecht. Proposals need to be submitted to the institutional ethical review board of the University Medical Center Utrecht. After review, the data selection will be provided to the researcher.
Supporting Information: Study Protocol, CSR
Time Frame: In view of the regulation for clinical trials, the investigators need to save all data for at least 15 years with the goal to be able to go back to patient level. After finishing the project all documents and data are stored at the UMC Utrecht.
Access Criteria: The data manager keeps the linking table to personal data.

REFERENCES:
- See also: Het knieregister: register voor kniebehandelingen — https://www.umcutrecht.nl/nl/ziekenhuis/wetenschappelijk-onderzoek/het-knieregister-register-voor-kniebehandelingen
- See also: Knee joint distraction in regular care for treatment of knee osteoarthritis: A comparison with clinical trial data. — https://www.ncbi.nlm.nih.gov/pubmed/31968005
- See also: ICRS Patient Registry — https://cartilage.org/society/icrs-patient-registry/
- See also: Reduction of pin tract infections during external fixation using cadexomer iodine — https://rdcu.be/b93rq